CLINICAL TRIAL: NCT02494362
Title: Tele-rehabilitation in the Home With Gaming as a Method of Improving Upper Extremity Function After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Tony Szturm, Associate Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2015
Record Dates: First submitted 2015-05-22; First posted 2015-07-10 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Stroke; Hemiplegia
Keywords: Hand exercises; Hand function; Computer based exercises; Therapeutic gaming
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Group (Experimental): Computer gaming hand exercise regimen.
  Interventions: Other: Computer gaming hand exercise regimen.

INTERVENTIONS:
Other: Computer gaming hand exercise regimen. — Computer gaming hand exercise regimen using common objects of daily life. The hand exercises are coupled with commercially available computer games and will be performed 30 minutes,four times per week for 12 weeks.

SUMMARY:
The purpose of the study is to determine whether a novel computer gaming hand exercise regimen would improve hand and arm function and be feasible in people with hemiplegia after Stroke affecting the hand.

DETAILED DESCRIPTION:
A novel computer gaming hand exercise regimen has been designed for people with hemiplegia after Stroke affecting the hand. The design allows a broad range of common objects of daily life to be seamlessly transformed into 'therapeutic' input devices by instrumenting with a small motion sense mouse. Based on individual abilities and treatment needs, objects are selected to train specific fine/ gross dexterous functions. The object manipulations (therapeutic exercises) are then used to control and play any commercially available computer game, making practice challenging and engaging.

The study is of twelve weeks duration comparing the computer gaming and conventional hand exercises in ten people with hemiplegia after Stroke affecting the hand. The investigators hypothesize that the game based exercises will improve hand function and will be feasible. A mixed-effect repeated measures analysis of variance will be conducted to test pre to post treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Time since stroke onset less than 1 year.
* Ability to actively extend at least 10 degrees at the Metacarpophalangeal and Interphalangeal joints and 10 degrees at the wrist. At least 30 degree of active flexion-extension at elbow and some active movements present at the shoulder joint.
* English speaking.
* No clinical evidence of cognitive impairment (screened by physician or therapist).
* Have a personal computer at home.
* Lives in Winnipeg.
* Able to provide informed consent.

Exclusion Criteria:

* Patients having excessive spasticity, pain or contractures in the more affected limb will not be included in the study.
* Convulsive seizures preventing adequate attention to task.
* Problem with vision.
* Aphasia.
* Apraxia.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor Function Test (Change is being assessed) | Baseline and 12 weeks

SECONDARY OUTCOMES:
Stroke Impact Scale (Change is being assessed) | Baseline and 12 weeks
Change from baseline in Paddle game based hand function assessment tool from baseline and 12 weeks. | Baseline and 12 weeks
  A novel, paddle game based hand function assessment tool has been developed designed to: 1) Objectively quantify the quality of finger hand movements (task performance) during manipulation of broad range of common objects independent of physical properties, anatomical requirements and task goal/context, 2) Track changes in finger hand function over time and 3) Aid in clinical decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szturm, PhD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - School of Medical Rehabilitation , University of Mantioba, Winnipeg, Manitoba
  - Riverview Health Centre, Winnipeg, Manitoba

REFERENCES:
- [Background] Szturm T, Peters JF, Otto C, Kapadia N, Desai A. Task-specific rehabilitation of finger-hand function using interactive computer gaming. Arch Phys Med Rehabil. 2008 Nov;89(11):2213-7. doi: 10.1016/j.apmr.2008.04.021. PMID 18996252
- [Background] Lockery D, Peters JF, Ramanna S, Shay BL, Szturm T. Store-and-feedforward adaptive gaming system for hand-finger motion tracking in telerehabilitation. IEEE Trans Inf Technol Biomed. 2011 May;15(3):467-73. doi: 10.1109/TITB.2011.2125976. PMID 21536526
- [Background] Andersen Hammond ER, Shay BL, Szturm T. Objective evaluation of fine motor manipulation-a new clinical tool. J Hand Ther. 2009 Jan-Mar;22(1):28-35; quiz 36. doi: 10.1197/j.jht.2008.06.006. Epub 2008 Aug 30. PMID 18950989